CLINICAL TRIAL: NCT02587949
Title: The Correlation Between Hair Cortisol Level of Acute Stroke or Its Long Term Disability.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0065-15-BNZ
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Cerebrovascular Stroke
Keywords: acute cerebrovascular stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In patients admitted to hospital with acute cerebrovascular stroke, we want to study the relationship between hair cortisol levels and biomarkers of inflammation and the clinical and radiological severity of the stroke and the degree of neurological disability being tested in three months and one year after.

DETAILED DESCRIPTION:
The study will include patients hospitalized due to an acute cerebrovascular stroke. A number of 30 patients aged 40-70 will be included. Within 48 hours of the event, blood inflammatory biomarkers, and scalp hair sample for cortisol will be taken. All recruited patients will undergo full neurological examination and the severity of the stroke will be rated using NIHSS (National Institutes of Health Stroke Scale). 3 months and one year later neurological examination and rating of neurological disability will be determined using Rankin Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 40-80.
2. Acute cerebrovascular stroke (symptoms that began no more than 72 hours before)
3. Rankin 0-1 before the event

Exclusion criteria:

1. Suspicion or known Cushing's syndrome
2. Known adrenal failure
3. Chronic inflammatory disease
4. Active malignancy
5. Acute infectious disease within 4 months before enrollment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients aged 40-80.
  2. Acute cerebrovascular stroke (symptoms that began no more than 72 hours before)
  3. Rankin 0-1 before the event
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Anti Tumor Necrosis Factor alpha | 24 months
  single blood sample will be drawn to measure Anti Tumor Necrosis Factor alpha levels (pg/ml).
C-reactive protein levels | 24 months
  single blood sample will be drawn to measure c-reactive protein levels (mcg/dl).
Hair Cortisol level | 24 months
  single hair sample will be drawn to measure cortisol levels (mcg/dl)
INL-6 | 24 months
  single blood sample will be drawn to measure INL-6 levels.

SECONDARY OUTCOMES:
TSH | 24 months
  single blood sample will be drawn to measure Thyroid-Stimulating Hormone (mcIU/ml).
FT4 | 24 months
  single blood sample will be drawn to measure Free Thyroxine (pmol/L) .
FT3 | 24 months
  single blood sample will be drawn to measure Free Triiodothyronine (pmol/L).
Cortisol | 24 months
  single blood sample will be drawn to measure cortisol levels (mcg/dl).

CONTACTS AND LOCATIONS:
Locations (1):
- Mira Koch, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided